CLINICAL TRIAL: NCT02994732
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-BVD-523 Following Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Absorption, Metabolism and Excretion (AME) of Single Dose Radiolabeled BVD-523 in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 523HV001
Record Dates: First submitted 2016-11-14; First posted 2016-12-16 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — ulixertinib

ARMS (1):
- [14C]-BVD-523 600mg single dose (Experimental): Open-label, nonrandomized, absorption, metabolism, and excretion study of [14C]-BVD-523 administered as a 600 mg (approximately 200 µCi) oral dose to 6 healthy male subjects following at least an 8-hour fast from food (not including water).
  Interventions: Drug: [14C]-BVD-523

INTERVENTIONS:
Drug: [14C]-BVD-523 — [14C]-BVD-523 administered as a 600-mg (approximately 200 µCi) oral dose to 6 healthy male subjects following a 2-hour fast from food (not including water) that follows breakfast.
  Other Names: Ulixertinib

SUMMARY:
The primary objective of this study is to characterize the metabolic disposition, pharmacokinetics (PK), and routes of elimination of [14C]-labeled BVD-523 after administration of a single, oral dose to healthy male subjects.

The secondary objective of this study is to evaluate the safety and tolerability of a single oral dose of [14C]-labeled BVD-523 in healthy male subjects.

DETAILED DESCRIPTION:
This study will be an open-label, absorption, metabolism, and excretion study of [14C]-BVD-523 administered as a 600-mg (approximately 200 µCi) oral dose to 6 healthy male subjects following a 2-hour fast from food (not including water) that follows breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Males, between 18 and 65 years of age, inclusive, at Screening
* Have a body mass index range of 18.5 to 32.0 kg/m2, inclusive, at Screening
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs measurements at Screening or Check-in and PE findings at Check-in as determined by the Investigator (or designee)
* Clinical laboratory evaluations (including clinical chemistry panel [fasted at least 8 hours], hematology/complete blood count [CBC], and urinalysis [UA] within the reference range for the test laboratory at Screening and Check-in, unless deemed not clinically significant by the Investigator (or designee)
* Negative test for selected drugs of abuse and cotinine at Screening (does not include alcohol) and at Check-in (does include alcohol)
* Negative hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody) and negative human immunodeficiency virus (HIV) antibody screens at Screening
* Males will be surgically sterile for at least 90 days (confirmed by documented azoospermia) or, when sexually-active with female partners of child-bearing potential, will agree to use contraception as detailed in Section 6.3.3 from Check-in until 90 days following Discharge
* Males must be willing to refrain from sperm donation from Check-in to 90 days from day of dosing
* Able to comprehend and willing to sign an ICF
* A minimum of 1 bowel movement per day.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, infectious, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator [or designee]) prior to Check-in
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) prior to Check-in
* History of stomach or intestinal surgery or resection that could alter absorption or excretion of orally administered drugs prior to Check-in except appendectomy, and hernia repair will be allowed if it was not associated with;
* History of Gilbert's Syndrome
* History or presence of an abnormal ECG that, in the Investigator's (or designee's) opinion, is clinically significant
* History of alcoholism or drug addiction within 1 year prior to Check-in
* History of nicotine use within 6 months prior to Check-in or positive cotinine at Screening or Check-in
* Participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in. The previous radiolabeled study drug must have been received more than 6 months prior to Check-in for this study and the total exposure from this study and the previous study will be within the recommended levels considered safe, per United States (US) Title 21 Code of Federal Regulations (CFR) 361.1 (eg, less than 3,000 mrem whole body annual exposure)
* Exposure to significant radiation (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to Check-in
* Use of any drugs or substances known to be strong inhibitors or strong inducers of CYP3A enzyme within 30 days prior to study drug administration, unless otherwise stated, and throughout the study
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days prior to Check-in, whichever is longer
* Use of any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee)
* Use of any over-the-counter, nonprescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee)
* Poor peripheral venous access prior to Check-in
* Donation of whole blood from 56 days prior to Screening through Discharge, inclusive, or of plasma from 30 days prior to Screening through Discharge, inclusive
* Receipt of blood products within 2 months prior to Check-in
* Any acute or chronic condition that, in the opinion of the Investigator (or designee), would limit the subject's ability to complete or participate in this clinical study
* Any other unspecified reason that, in the opinion of the Investigator (or designee) or Sponsor, make the subject unsuitable for enrollment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Covance

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental [14C] - BVD-523 600mg Single Dose: Subjects received a single oral 600-mg (4 ×150-mg capsules) dose of BVD-523 containing approximately 200 µCi of [14C] labeled BVD-523 following a 2-hour fast that followed breakfast. Six subjects were enrolled in, dosed, and completed study. All six subjects were male, 4 subjects were white and 2 subjects were black or African American.
Period: Overall Study
Arm/Group | Experimental [14C] - BVD-523 600mg Single Dose
Started | 6 (All subjects entered clinic on January 11, 2017)
Completed | 6 (All subjects were discharged from the clinic by Jan 24, 2017)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study: Six subjects were enrolled in, dosed, and completed study. All six subjects were male, 4 subjects were white and 2 subjects were black or African American.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.9 (2.38)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of 14C-labeled BVD-523(Radioactivity in Whole Blood and Plasma) Tmax
Description: Time to peak concentration (Tmax), PK blood samples were taken at the following time points 0 (predose), 30 min, 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post dose.
Time Frame: Collected over 5 days
Population: All enrolled subjects
Measure: Median (Standard Deviation); unit: hr
Groups:
- Experimental [14C] -BVD-523 600mg Single Dose: Subjects will receive a single oral 600-mg (4 ×150-mg capsules) dose of BVD-523 containing approximately 200 µCi of [14C] labeled BVD-523 following a 2-hour fast that follows breakfast. Six subjects were enrolled in, dosed, and completed study. All six subjects were male, 4 subjects were white and 2 subjects were black or African American.
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
hr | 2.57 (3.0)

2. Primary Outcome: Pharmacokinetics of 14C-labeled BVD-523(Radioactivity in Whole Blood and Plasma) Cmax
Description: peak (maximum) concentration
Time Frame: Collected over 5 days
Population: All 6 subjects enrolled
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
ng/ml | 1110 (619)

3. Primary Outcome: Pharmacokinetics of 14C-labeled BVD-523(Radioactivity in Whole Blood and Plasma) t1/2
Description: Elimination half-life
Time Frame: Collected over 15 days
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
hr | 8.75 (3.57)

4. Primary Outcome: Pharmacokinetics of 14C-labeled BVD-523(Radioactivity in Whole Blood and Plasma) AUC
Description: Area under Curve (AUC), 0-24 hr
Time Frame: Collected over 15 dyas
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
hr*ng/ml | 8480 (3600)

5. Primary Outcome: Pharmacokinetics of 14C-labeled BVD-523(Radioactivity in Whole Blood and Plasma) CL/F
Description: Oral Clearance (CL/F)
Time Frame: Collected over 15 days
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
L/hr | 73 (35.1)

6. Primary Outcome: Pharmacokinetics of 14C-labeled BVD-523(Radioactivity in Whole Blood and Plasma) V/F
Description: Apparent volume of distribution (V/F)
Time Frame: Collected over 15 days
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
L | 899 (463)

7. Primary Outcome: Excretion Rate of 14C-labeled BVD-523(Radioactivity in Feces)
Description: Percent of dose excreted in feces
Time Frame: Collected over 15 days
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: %of radioactive dose of [14C-BVD523
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
%of radioactive dose of [14C-BVD523 | 82 (4.72)

8. Primary Outcome: Excretion Rate of 14C-labeled BVD-523(Radioactivity in Urine)
Description: Percent of dose excreted in urine
Time Frame: Collected over 15 days
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: % of radioactive dose of [14C-BVD523
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
% of radioactive dose of [14C-BVD523 | 14.8 (4.79)

9. Primary Outcome: Cumulative Whole Blood: Plasma Ratio Calculated for AUC0-12
Description: AUC from time zero to the 12 hr time point with concentration above the lower limit of quantitation
Time Frame: Collected in 12 hrs
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
hr*ng/ml | 0.464 (0.0354)

10. Primary Outcome: Cumulative Whole Blood: Plasma Ratio Calculated for AUC 0-24
Description: AUC from time zero to 24 hrs
Time Frame: Collected in 24 hrs
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Experimental [14C] -BVD-523 600mg Single Dose
Number analyzed (Participants) | 6
hr*ng/ml | 0.409 (0.0297)

11. Secondary Outcome: Treatment-related Adverse Events
Description: Any treatment-emergent adverse events related or likely related to study treatment
Time Frame: 27 days
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
Participants | 2

ADVERSE EVENTS:
Time Frame: 27 days
Description: Adverse event definitions; assignment of severity, causality, action taken, and outcome; and procedures for reporting serious AEs (SAEs) are detailed in Appendix C of the protocol. None of the definitions differ from the clinicaltrials.gov definitions.
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=6)
Fatigue (General disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT02994732/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT02994732/SAP_001.pdf